CLINICAL TRIAL: NCT02718053
Title: Reliability of Spasticity Measurement With Lokomat
Status: Suspended | Type: Observational
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Principal Investigator, Ilaria Zivi, MD, Ospedale Generale Di Zona Moriggia-Pelascini
Other Study IDs: spasticity01
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Spasticity, Lokomat
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- spasticity: patients affected by spasticity of the lower limbs
  Interventions: Other: L-stiff; Other: Ashworth
- controls: healthy subjects
  Interventions: Other: L-stiff; Other: Ashworth

INTERVENTIONS:
Other: L-stiff — spasticity measurement with Lokomat
Other: Ashworth — spasticity measurement with Ashworth scale

SUMMARY:
The purpose of the study is to evaluate the reliability of spasticity measurement with Lokomat

ELIGIBILITY:
Inclusion Criteria:

* patients affected by lower limbs spasticity

Exclusion Criteria:

* medical contraindications to mobilization with Lokomat

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: subjects are selected from patients hospitalized in our neurorehabilitation unit
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
correlation of spasticity measurement obtained with L-Stiff (Lokomat) and Ashworth scale | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Generale di Zona Moriggia Pelascini, Gravedona Ed Uniti, CO, Italy